CLINICAL TRIAL: NCT00666692
Title: Phase 1b Trial Evaluating the Safety of Volociximab in Combination With Carboplatin, Paclitaxel, and Bevacizumab in Subjects With Previously Untreated Stage IIIB/IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Phase 1b Study With Volociximab in Combination With Carboplatin, Paclitaxel, and Bevacizumab in First-line, Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M200-1212
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cancer; carcinoma; monoclonal antibody therapy; anti-angiogenesis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Carcinoma | interventions — volociximab; Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Escalating doses of volociximab at 10, 20, and 30 mg/kg with carboplatin, paclitaxel, and bevacizumab
  Interventions: Drug: M200 (Volociximab), Carboplatin, Paclitaxel, Bevacizumab

INTERVENTIONS:
Drug: M200 (Volociximab), Carboplatin, Paclitaxel, Bevacizumab — Volociximab will be administered via IV infusion once every three week at 10, 20, and 15 or 30 mg/kg with an additional loading dose in the 10, 20, and 15 mg/kg dose levels on Day 8 of the first cycle. Volociximab will be given for up to 6 cycles (3 weeks/cycle). Subjects who have stable disease or better and subjects who have disease that is not progressing at the end of 6 cycles may continue to receive volociximab alone until disease progression. Carboplatin is administered via IV infusion and dosed based on the Calvert formula (with a target area AUC of 6 mg/mL/min) for up to 6 cycles (3 weeks/cycle). Paclitaxel is administered via IV infusion and dosed at 200 mg/m2 for up to 6 cycles (3 weeks/cycle). All four drugs, when given in combination, will be infused on the same day in the following sequence: volociximab, paclitaxel, carboplatin.
  Other Names: Volociximab (M200)

SUMMARY:
The primary purpose of this study is to examine the safety of volociximab (V) in combination with a standard treatment of carboplatin (C), paclitaxel (P), and bevacizumab (B) in subjects previously untreated with chemotherapy for advanced stage (IIIB/IV) non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Phase 1b, multicenter, open-label, dose-escalation study to evaluate the safety and tolerability of volociximab in combination with C/P + B in subjects with previously untreated Stage IIIB/IV non-squamous NSCLC.

Subjects will be treated with the C/P + B + volociximab (V)combination for a total of 6 cycles (3 weeks/cycle). Subjects with stable disease (SD)or better per Response Evaluation Criteria in Solid Tumors (RECIST)after the 6th cycle of combination treatment (C/P + B + V) will be considered for further treatment in a maintenance phase with B + V at the same dose until subject withdrawal from treatment.

Volociximab will be administered at doses ranging from 10 to 30 mg/kg every 3 weeks. Paclitaxel, carboplatin, and bevacizumab will be administered at their registered doses for this combination.

Follow up for each subject will extend over a 90-day period following the last dose of volociximab. End of study is defined as 90 days after the last dose of volociximab for the last subject treated in the study.

ELIGIBILITY:
Inclusion Criteria

* Males and females of at least 18 years of age.
* Stage IIIB with pleural effusion or Stage IV non-squamous NSCLC.
* Measurable and/or evaluable disease according to RECIST.
* No prior chemotherapy, biological therapy or immunotherapy for Stage IIIB/IV disease. Adjuvant therapy for early stage disease must have been completed > or = 6 months prior to Cycle 1, Day 1 of this study.
* Eastern Cooperative Oncology Group (ECOG) performance status < or =1.
* A negative pregnancy test (serum or urine) in women of childbearing potential at screening. Male subjects and female subjects of childbearing potential must be willing to practice effective contraception during the study and be willing and able to continue contraception for 6 months after the last dose of study drug.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) (in accordance with national and local subject privacy regulations).

Exclusion Criteria

* Histological evidence of predominantly squamous cell carcinoma.
* Known central nervous system (CNS) metastases.
* Known allergy or sensitivity to murine proteins, chimeric antibodies or other components of the product, Cremophor EL (polyoxyethylated castor oil), cisplatin, or other platinum-containing compounds.
* Absolute neutrophil count (ANC) <1500/mm3, hemoglobin level <10 g/dL, or a platelet count <100,000/mm3.
* Aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase values of .2.5 of the upper limits of normal values (ULN) (>5 ULN for subjects with liver metastases) or alkaline phosphatase values >2.5 ULN (unless documented bone metastases are responsible for the increase of alkaline phosphatase); total bilirubin >1.5 mg/dL, or serum creatinine >1.8 mg/dL.
* Radiation therapy within 1 month before Cycle 1, Day 1.
* Documented symptomatic central nervous system (CNS) tumor or CNS metastases.
* History of thromboembolic events, including cardiovascular or cerebrovascular events (ie, acute myocardial infarction [AMI], stroke) within 1 year prior to Cycle 1, Day 1.
* History of known bleeding disorders and coagulation defects.
* History of significant hemoptysis (ie, > or = 1/2 teaspoon red blood per event) or gastrointestinal bleeding within 1 year prior to Cycle 1, Day 1.
* Major surgery (eg, exploratory laparotomy) within 4 weeks prior to Cycle 1, Day 1 of the study.
* Clinically significant or unstable medical conditions including, but not limited to, uncontrolled diabetes mellitus requiring insulin, uncontrolled hypertension, or uncontrolled or symptomatic orthostatic hypotension.
* Oxygen-dependent chronic obstructive pulmonary disease.
* Known active infections requiring intravenous (IV) antibiotics, antivirals, or antifungals, including but not limited to chronic human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Prior bone marrow or stem cell transplant.
* Regular use of aspirin, nonsteroidal anti-inflammatory agents, or other agents known to inhibit platelet function.
* High-dose warfarin or heparin use. [Note: Low-dose warfarin (1 mg/day) or low-dose heparin for IV-catheter patency, and low-molecular weight heparin for prophylaxis are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of volociximab given at different doses in combination with carboplatin, paclitaxel, and bevacizumab. | Dose Limiting Toxicities (DLT) will be assessed during the first treatment cycle for each cohort

SECONDARY OUTCOMES:
1) Pharmacokinetics of volociximab 2) Efficacy of volociximab in combination with carboplatin/paclitaxel and bevacizumab. | Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — Abbott
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 70354, Bethesda, Maryland
  - Site Reference ID/Investigator# 70333, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 70355, Greenville, South Carolina
  - Site Reference ID/Investigator# 70353, Yakima, Washington